# Opioid-Free Anesthesia vs Opioid-Based Anesthesia in Laparoscopic Bariatric Surgery

NCT Number: NCTXXXXXXX

Document Date: 01 July 2023

#### Title

Opioid-Free Anesthesia vs Opioid-Based Anesthesia in Laparoscopic Bariatric Surgery

#### Version

1.0

# **Principal Investigator**

Emanuel Almeida, MD, Consultant Anesthesiologist

Institution: Hospital Lusíadas Amadora – Lusíadas Saúde, S.A.

# 1. Background and Rationale

Obesity is a chronic disease commonly associated with complications. Bariatric surgery is effective, but pain and PONV remain challenges. Opioid-free anesthesia (OFA) may reduce opioid-related adverse effects. This trial compares OFA vs. OBA in laparoscopic bariatric surgery.

# 2. Objectives

Primary: Compare postoperative pain (NRS) between OFA and OBA.

Secondary: NOL index; rescue analgesia; opioid consumption; PONV; satisfaction; complications; LOS.

# 3. Study Design

Interventional, prospective, randomized, parallel-group clinical trial.

Allocation: Randomized

Masking: None (open-label)

Arms: 2

Primary Purpose: Treatment

Phase: Not applicable

## 4. Study Arms and Interventions

Arm 1 – OBA: Remifentanil infusion; propofol; rocuronium; desflurane; dexamethasone; cefazolin; esomeprazole; postoperative multimodal analgesia; rescue opioids.

Arm 2 – OFA: Dexmedetomidine bolus + infusion with ketamine and lidocaine; propofol; rocuronium; desflurane; postoperative opioid-free analgesia; rescue tramadol.

## 5. Eligibility Criteria

Inclusion: Adults  $\geq$ 18 years; BMI  $\geq$ 35 with comorbidities or  $\geq$ 40; elective laparoscopic bariatric surgery; consent.

Exclusion: Pregnancy; substance abuse; severe psychiatric disease; contraindication to study drugs.

#### 6. Outcomes

Primary: Postoperative pain (NRS) at PACU arrival, PACU discharge, 24h, discharge.

Secondary: NOL index; rescue analgesia; opioid consumption; PONV; satisfaction; complications; LOS.

# 7. Sample Size

60 participants (30 per arm). Convenience sample based on feasibility.

### 8. Randomization

Computer-generated 1:1 allocation.

## 9. Blinding

None (open-label).

### 10. Data Collection

NRS, PONV, rescue analgesia, satisfaction, complications; NOL intraoperative at multiple time points.

## 11. Statistical Analysis

Shapiro–Wilk; t-test; Mann–Whitney; chi-square; GLM with Bonferroni; significance p < 0.05.

### 12. Ethical Considerations

Approved by the Ethics Committee of Hospital Lusíadas Amadora. Written informed consent obtained.

### 13. Data Management

Password-protected storage. No IPD sharing.

#### 14. Dissemination Plan

Results will be published in peer-reviewed journals.

#### 15. Timeline

Start, end, and completion dates to be added.